CLINICAL TRIAL: NCT00080223
Title: An Open-Label, Phase 2 Study of the Safety of Oral Pirfenidone in Patients With Pulmonary Fibrosis/Idiopathic Pulmonary Fibrosis
Brief Title: Safety Study of Oral Pirfenidone in Patients With Pulmonary Fibrosis/Idiopathic Pulmonary Fibrosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PIPF-002; GA29989 (Other: Hoffmann-La Roche)
Record Dates: First submitted 2004-03-24; First posted 2004-03-26 (Estimated); Results first posted 2016-03-09 (Estimated); Last update posted 2017-04-17 (Actual); Status verified 2017-03

CONDITIONS: Idiopathic Pulmonary Fibrosis; Pulmonary Fibrosis
Keywords: pulmonary fibrosis; respiratory diseases
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Pulmonary Fibrosis; Respiratory Tract Diseases | interventions — pirfenidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pirfenidone (Experimental): up to 3600 mg/day of pirfenidone given orally administered in divided doses three times daily with food, for the duration of the study
  Interventions: Drug: Pirfenidone

INTERVENTIONS:
Drug: Pirfenidone — up to 3600 mg/day of pirfenidone given orally administered in divided doses three times daily with food, for the duration of the study

SUMMARY:
To assess the safety of treatment with pirfenidone (up to 3600 mg/d) in patients with pulmonary fibrosis/idiopathic pulmonary fibrosis (PF/IPF).

DETAILED DESCRIPTION:
This study has been designed as a rollover study to collectively include safety data from various previous studies.

In addition, InterMune has also initiated an Early Access Program to make pirfenidone available to a limited number of patients with idiopathic pulmonary fibrosis in the United States. This program is also being conducted under this protocol. Registration of patients with documented IPF has been closed as of October 2005.

ELIGIBILITY:
General Inclusion Criteria:

* Able to understand and sign an informed consent form
* Understand the importance of adherence to study treatment and the study protocol, including concomitant medication restrictions, throughout the study period
* Patients must be willing to travel to an approved regional center for all study-related visits

Roll-Over Criteria:

* Entry into study through rollover has been completed

Criteria for Early Access Program patients:

* Clinical symptoms consistent with IPF ≥3 months duration
* Age 40 - 85, inclusive
* At the time of registration with National Organization for Rare Disorders (NORD), patients with IPF must have a percent predicted forced vital capacity (FVC) of ≥50%, and percent predicted carbon monoxide diffusing capacity (DLCO) of ≥35%
* At the time of enrollment in PIPF-002, (screening/baseline visit) percent predicted FVC must be ≥45%, and percent predicted DLCO must be ≥30%
* High-resolution computed tomographic scan (HRCT) showing definite IPF. For patients with surgical lung biopsy showing definite or probable usual interstitial pneumonia (UIP), the HRCT criterion of probable IPF is sufficient
* For patients aged <50 years: open or video-assisted thoracoscopic (VATS) lung biopsy showing definite or probable UIP. In addition, no features supporting an alternative diagnosis on transbronchial biopsy or bronchoalveolar lavage if performed
* For patients aged ≥50 years: at least one of the following diagnostic findings as well as the absence of any features on specimens resulting from any of these procedures that support an alternative diagnosis: 1) Open or VATS lung biopsy showing definite or probable UIP; 2) Transbronchial biopsy showing no features to support an alternative diagnosis; 3) Bronchoalveolar lavage (BAL) showing no features to support an alternative diagnosis

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2003-08-31 (Actual); Primary Completion 2015-04-30 (Actual); Study Completion 2015-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (25):
- United States (25):
  - Phoenix, Arizona
  - Pomona, California
  - San Jose, California
  - New Haven, Connecticut
  - Sarasota, Florida
  - Atlanta, Georgia
  - Kailua, Hawaii
  - Lahaina, Hawaii
  - Nampa, Idaho
  - Elk Grove Village, Illinois
  - Boston, Massachusetts
  - West Roxbury, Massachusetts
  - St Louis, Missouri
  - Huntington Station, New York
  - New York, New York
  - Rochester, New York
  - Worthington, Ohio
  - Portland, Oregon
  - Lancaster, Pennsylvania
  - Dallas, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Provo, Utah
  - Annandale, Virginia
  - Bremerton, Washington

REFERENCES:
- [Derived] Gotfried MH, Girod CE, Antin-Ozerkis D, Burgess T, Strombom I, Stauffer JL, Kirchgaessler KU, Padilla ML. An Open-Label, Phase II Study of the Safety of Pirfenidone in Patients with Idiopathic Pulmonary Fibrosis (PIPF-002). Pulm Ther. 2018 Jun;4(1):59-71. doi: 10.1007/s41030-018-0053-y. Epub 2018 Apr 5. PMID 32026243

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants could enroll from Study PIPF-001 (a double-blind comparison of pirfenidone and prednisone in pulmonary fibrosis); individual-patient protocols (IPPs); investigator-sponsored Investigational New Drug applications (INDs) in idiopathic pulmonary fibrosis (IPF); and via an early access program (EAP) for participants with IPF.
Groups:
- Pirfenidone: Pirfenidone was administered orally, in divided doses, three times daily at a maximum dose of up to 3600 milligram per day (mg/d). At the start of treatment in this study, doses for participants with no previous pirfenidone exposure and for those who took their last dose greater than (>) 4 weeks before enrollment were titrated to their maintenance dose based on body weight and tolerability. Dose titration was also required after a dosing interruption of >28 days. Pirfenidone was administered for a maximum duration of 604 weeks in this study.
Period: Overall Study
Arm/Group | Pirfenidone
Started | 83
Completed | 7
Not Completed | 76
Not completed — Adverse Event | 23
Not completed — Death | 21
Not completed — Withdrawal by Subject | 13
Not completed — Lung Transplantation | 9
Not completed — Non-compliance With Study Treatment | 7
Not completed — Participant unwilling to continue | 2
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Population: All treated participants
Groups:
- Pirfenidone: Pirfenidone was administered orally, in divided doses, three times daily at a maximum dose of up to 3600 mg/d. At the start of treatment in this study, doses for participants with no previous pirfenidone exposure and for those who took their last dose >4 weeks before enrollment were titrated to their maintenance dose based on body weight and tolerability. Dose titration was also required after a dosing interruption of >28 days. Pirfenidone was administered for a maximum duration of 604 weeks in this study.
Arm/Group | Pirfenidone
Number analyzed (Participants) | 83
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.5 (9.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 60

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Treatment-Emergent Adverse Event (AE), Serious AE (SAE), Severe AE, Life-threatening AE, Death or Discontinuation Because of an AE
Description: An AE was any untoward medical occurrence attributed to study drug in a participant who received study drug. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. AEs were classified as severe (Grade 3) in following cases: marked limitation in activity; some assistance usually required; medical intervention/ therapy required, hospitalization possible. Treatment-emergent AEs were those occurring on or after the first dosing day and up to 28 days after discontinuation of study treatment, and those occurring before treatment that worsened after the first study dose. AE included serious as well as non-serious AEs.
Time Frame: Baseline to 28 days after the last dose of study treatment (maximum duration of treatment in study was 604 weeks)
Population: All treated participants
Measure: Number; unit: percentage of participants
Arm/Group | Pirfenidone
Number analyzed (Participants) | 83
percentage of participants
  Any AE | 98.8
  SAE | 59.0
  Severe AE | 36.1
  Life-threatening AE | 21.7
  AEs leading to death | 25.3
  AE leading to study treatment discontinuation | 43.4

2. Secondary Outcome: Percent Predicted Forced Vital Capacity (FVC)
Description: FVC is a standard pulmonary function test used to quantify respiratory muscle weakness. FVC is the volume of air that can forcibly be blown out from the lungs after full inspiration in the upright position, measured in liters. Predicted FVC is based on a formula using sex, age and height of a person, and is an estimate of healthy lung capacity. Percent of predicted FVC = (actual FVC value in liter)/(predicted FVC) * 100%
Time Frame: Baseline, Weeks 24, 48, 72, 96, 120, 144, 168, 192, 216, 240, 264, 288, 312, 336, 360, 384, 408, 432, 456, 480
Population: All treated participants. "n" = participants who were evaluable for specified time point.
Measure: Mean (Standard Deviation); unit: percent predicted FVC
Arm/Group | Pirfenidone
Number analyzed (Participants) | 83
percent predicted FVC
  Baseline (n=78) | 67.7 (18.70)
  Week 24 (n=71) | 67.5 (17.11)
  Week 48 (n=57) | 68.7 (17.36)
  Week 72 (n=50) | 68.4 (16.20)
  Week 96 (n=47) | 67.9 (17.76)
  Week 120 (n=44) | 67.7 (18.03)
  Week 144 (n=39) | 66.1 (18.22)
  Week 168 (n=35) | 65.7 (17.74)
  Week 192 (n=28) | 67.8 (18.32)
  Week 216 (n=28) | 68.7 (21.97)
  Week 240 (n=22) | 65.3 (16.80)
  Week 264 (n=15) | 70.1 (13.26)
  Week 288 (n=14) | 76.6 (18.71)
  Week 312 (n=14) | 71.1 (14.03)
  Week 336 (n=10) | 64.9 (13.61)
  Week 360 (n=7) | 60.9 (15.00)
  Week 384 (n=6) | 68.4 (17.43)
  Week 408 (n=4) | 65.1 (11.84)
  Week 432 (n=1) | 61.5 (NA) — Standard deviation was not available as there was only 1 participant analyzed for this time point.
  Week 456 (n=1) | 78.4 (NA) — Standard deviation was not available as there was only 1 participant analyzed for this time point.
  Week 480 (n=1) | 80.9 (NA) — Standard deviation was not available as there was only 1 participant analyzed for this time point.

3. Secondary Outcome: Hemoglobin (Hgb)-Corrected Percent-Predicted Carbon Monoxide Diffusing Capacity (DLco)
Description: DLco is a pulmonary function test, and measures the partial pressure difference between inspired and expired carbon monoxide. Predicted DLco is based on a formula using sex, age and height of a person. Predicted DLco = [Hbg-corrected DLco value (in milliliters per minute per millimeter mercury [mL/min/mmHg])/predicted DLco] * 100%
Time Frame: Baseline, Weeks 24, 48, 72, 96, 120, 144, 168, 192, 216, 240, 264, 288, 312, 336, 360, 384, 408, 432, 456, 480
Population: All treated participants. "n" = participants who were evaluable for specified time point.
Measure: Mean (Standard Deviation); unit: percent predicted DLco
Arm/Group | Pirfenidone
Number analyzed (Participants) | 83
percent predicted DLco
  Baseline (n=74) | 38.0 (13.36)
  Week 24 (n=65) | 39.5 (13.56)
  Week 48 (n=55) | 37.1 (13.55)
  Week 72 (n=49) | 37.0 (12.01)
  Week 96 (n=44) | 38.0 (12.35)
  Week 120 (n=41) | 35.7 (12.55)
  Week 144 (n=37) | 38.5 (13.47)
  Week 168 (n=33) | 36.7 (12.98)
  Week 192 (n=27) | 37.2 (11.34)
  Week 216 (n=28) | 35.8 (11.31)
  Week 240 (n=22) | 35.5 (12.67)
  Week 264 (n=15) | 37.5 (9.69)
  Week 288 (n=14) | 42.9 (18.43)
  Week 312 (n=14) | 38.6 (9.54)
  Week 336 (n=10) | 33.7 (6.41)
  Week 360 (n=7) | 37.1 (11.19)
  Week 384 (n=5) | 38.3 (13.16)
  Week 408 (n=4) | 38.1 (9.41)
  Week 432 (n=1) | 33.9 (NA) — Standard deviation was not available as there was only 1 participant analyzed for this time point.
  Week 456 (n=1) | 11.6 (NA) — Standard deviation was not available as there was only 1 participant analyzed for this time point.
  Week 480 (n=1) | 38.9 (NA) — Standard deviation was not available as there was only 1 participant analyzed for this time point.

4. Secondary Outcome: Resting Oxygen Saturation by Pulse Oximetry (SpO2)
Description: SpO2 is the percentage of oxygen saturation in the blood. Oxygen level (oxygen saturation) of the blood was measured using pulse oximetry on room air.
Time Frame: Baseline, Weeks 24, 48, 72, 96, 120, 144, 168, 192, 216, 240, 264, 288, 312, 336, 360, 384, 408, 432, 456, 480
Population: All treated participants. "n" = participants who were evaluable for specified time point.
Measure: Mean (Standard Deviation); unit: percentage of oxygen saturation
Arm/Group | Pirfenidone
Number analyzed (Participants) | 83
percentage of oxygen saturation
  Baseline (n=72) | 94.5 (3.53)
  Week 24 (n=55) | 94.4 (4.14)
  Week 48 (n=47) | 94.8 (3.05)
  Week 72 (n=41) | 94.9 (3.01)
  Week 96 (n=36) | 94.9 (2.77)
  Week 120 (n=35) | 94.8 (2.46)
  Week 144 (n=33) | 94.8 (2.78)
  Week 168 (n=25) | 94.0 (3.18)
  Week 192 (n=22) | 94.9 (2.59)
  Week 216 (n=23) | 95.2 (2.33)
  Week 240 (n=17) | 95.5 (2.67)
  Week 264 (n=11) | 95.7 (1.56)
  Week 288 (n=10) | 94.6 (4.09)
  Week 312 (n=11) | 95.8 (2.48)
  Week 336 (n=9) | 94.4 (2.35)
  Week 360 (n=7) | 94.9 (4.02)
  Week 384 (n=7) | 94.0 (2.77)
  Week 408 (n=6) | 94.8 (2.86)
  Week 432 (n=1) | 95.0 (NA) — Standard deviation was not available as there was only 1 participant analyzed for this time point.
  Week 456 (n=1) | 97.0 (NA) — Standard deviation was not available as there was only 1 participant analyzed for this time point.
  Week 480 (n=3) | 95.0 (2.00)

5. Secondary Outcome: Overall Survival
Description: Survival was analyzed as time from first study dose to death (all-cause mortality) with surviving participants censored at their last available assessment.
Time Frame: First dosing of study treatment until death (up to 604 weeks)
Population: All treated participants
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Pirfenidone
Number analyzed (Participants) | 83
weeks | 508.7 [264.14 to NA] — The upper limit of the 95% confidence interval was not calculable because of higher (>50%) number of censored participants.

ADVERSE EVENTS:
Time Frame: Baseline to 28 days after the last dose of study treatment (maximum duration of treatment in study was 604 weeks)
Description: All treated participants
Arm/Group | Pirfenidone
Serious Adverse Events (participants affected / at risk) | 49/83
Other Adverse Events (participants affected / at risk) | 81/83
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pirfenidone (N=83)
Anaemia (Blood and lymphatic system disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 1
Angina pectoris (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 4
Atrial flutter (Cardiac disorders) | 1
Cardiac arrest (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 2
Coronary artery disease (Cardiac disorders) | 3
Coronary artery occlusion (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 2
Supraventricular tachycardia (Cardiac disorders) | 1
Ventricular fibrillation (Cardiac disorders) | 1
Abdominal hernia (Gastrointestinal disorders) | 1
Abdominal strangulated hernia (Gastrointestinal disorders) | 1
Colitis ischaemic (Gastrointestinal disorders) | 2
Diverticulum (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Oesophageal disorder (Gastrointestinal disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Bronchitis (Infections and infestations) | 3
Device related infection (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Lobar pneumonia (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 9
Respiratory tract infection (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Viral infection (Infections and infestations) | 1
Chest injury (Injury, poisoning and procedural complications) | 1
Facial bones fracture (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 1
Hip fracture (Injury, poisoning and procedural complications) | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1
Limb injury (Injury, poisoning and procedural complications) | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 1
Radius fracture (Injury, poisoning and procedural complications) | 1
Ulna fracture (Injury, poisoning and procedural complications) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Starvation (Metabolism and nutrition disorders) | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung squamous cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Autonomic nervous system imbalance (Nervous system disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 2
Dementia (Nervous system disorders) | 1
Encephalopathy (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Renal failure acute (Renal and urinary disorders) | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 15
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 6
Shock (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pirfenidone (N=83)
Anaemia (Blood and lymphatic system disorders) | 5
Abdominal discomfort (Gastrointestinal disorders) | 7
Constipation (Gastrointestinal disorders) | 10
Diarrhoea (Gastrointestinal disorders) | 10
Dyspepsia (Gastrointestinal disorders) | 7
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 10
Nausea (Gastrointestinal disorders) | 40
Stomach discomfort (Gastrointestinal disorders) | 5
Vomiting (Gastrointestinal disorders) | 13
Asthenia (General disorders) | 8
Fatigue (General disorders) | 27
Oedema peripheral (General disorders) | 9
Pyrexia (General disorders) | 7
Bronchitis (Infections and infestations) | 12
Nasopharyngitis (Infections and infestations) | 8
Respiratory tract infection (Infections and infestations) | 6
Sinusitis (Infections and infestations) | 11
Upper respiratory tract infection (Infections and infestations) | 21
Urinary tract infection (Infections and infestations) | 11
Contusion (Injury, poisoning and procedural complications) | 6
Skin laceration (Injury, poisoning and procedural complications) | 6
Weight decreased (Investigations) | 18
Anorexia (Metabolism and nutrition disorders) | 11
Decreased appetite (Metabolism and nutrition disorders) | 14
Back pain (Musculoskeletal and connective tissue disorders) | 10
Myalgia (Musculoskeletal and connective tissue disorders) | 6
Dizziness (Nervous system disorders) | 12
Headache (Nervous system disorders) | 14
Anxiety (Psychiatric disorders) | 10
Depression (Psychiatric disorders) | 12
Insomnia (Psychiatric disorders) | 15
Proteinuria (Renal and urinary disorders) | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 21
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 23
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 21
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 8
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 10
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 6
Pruritus (Skin and subcutaneous tissue disorders) | 5
Rash (Skin and subcutaneous tissue disorders) | 16
Hypertension (Vascular disorders) | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.